CLINICAL TRIAL: NCT00426413
Title: Ketosis Prone Diabetes Mellitus in African-Americans: Insulin Signaling, Proteomics, and Outcomes
Brief Title: Ketosis Prone Diabetes in African-Americans
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Dawn Smiley MD, Principal Investigator, Emory University
Other Study IDs: IRB00024857; GCRC 1703 (Other: Other); 897-2003 (Other: Other)
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Ketosis Prone Diabetes; Diabetic Ketoacidosis; Severe Hyperglycemia
Keywords: ketosis-prone diabetes; diabetic ketoacidosis; obesity; insulin dependence; mechanisms
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis; Hyperglycemia; Obesity | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study has IRB approval for blood sample collection for future DNA analyses and HLA typing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Obese AA subjects with DKA or severe hyperglycemia
  Interventions: Drug: pioglitazone
- 2: obese nondiabetic subjects, age 19-65.
- 3: Any subjects with recurrent DKA. Recurrent DKA is defined as more than one admission to Grady Memorial Hospital.

INTERVENTIONS:
Drug: pioglitazone — Obese AA subjects with DKA or severe hyperglycemia that are able to discontinue insulin at 12 weeks or less will be randomized (blinded fashion) to receive either placebo or pioglitazone qd. The subjects will be followed while in the study arm and beta-cell function will be assessed using OGTT at set intervals.
  Other Names: Actos (pioglitazone)
  Groups: 1

SUMMARY:
Over 50% of obese African-Americans (AA) presenting with newly diagnosed, severe hyperglycemia and/or unprovoked diabetic ketoacidosis (DKA) display clinical, metabolic, and immunogenetic features of type 2 diabetes. Prior studies indicate that these patients a) have markedly decreased insulin secretion and impaired insulin action at presentation, b) absent or low prevalence of beta-cell autoantibodies and c) are able to discontinue aggressive insulin therapy in ~70% of cases within 3 months of follow-up. These patients have been referred to as having ketosis-prone type 2 diabetes (KPDM). Most patients with KPDM, however, experience a hyperglycemic relapse within a year of insulin discontinuation. Consequently, patients with "KPDM" are an ideal model to follow throughout their clinical course. The specific aims of this proposal are to 1) identify clinical, metabolic, and immunogenetic markers that alone, or in combination, are predictive of short- and long-term near-normoglycemic remission and 2) determine whether pioglitazone or sitagliptin therapy will delay an insulin-deficient relapse once insulin is discontinued. The Principal Investigator hypothesizes that measures of beta-cell function at presentation, alone or in combination with measures of insulin sensitivity, will correlate with the ability of a patient to achieve and remain in near-normoglycemic remission. She also hypothesizes that intervention compared to placebo will preserve beta-cell function, improve insulin sensitivity, and prevent an insulin-deficient relapse. This prospective, cohort study with a RCT arm would better characterize the natural history of KPDM, facilitate the direction of long-term therapy, and likely decrease the recurrence of DKA which is associated with increased mortality and morbidity.

DETAILED DESCRIPTION:
More than half of obese African-Americans (AA) with newly diagnosed diabetes presenting with diabetic ketoacidosis (DKA) display clinical, metabolic, and immunogenetic features of type 2 diabetes during follow-up. Prior studies by our group and other investigators indicate that, at presentation, these patients a) have markedly decreased insulin secretion and impaired insulin action, b) have low prevalence of positive B-cell autoantibodies, and c) respond to aggressive diabetic management with significant improvement in B-cell function and insulin sensitivity sufficient to allow discontinuation of insulin therapy. Upon discontinuation of insulin, the period of near-normoglycemia remission (defined as the ability to discontinue insulin injections for ≥ one week and remain in good metabolic control - fasting blood glucose ≤ 120 mg/dl and A1c ≤ 7%) may last for a few months to several years. These patients are referred to as having atypical diabetes, Flatbush diabetes, or ketosis-prone type 2 diabetes (KPDM). Patients with "KPDM" are therefore an ideal model to follow throughout their clinical course in order to correlate their response to treatment with the mechanism(s) and markers of short- and long-term remission and determine the optimal therapeutic approach in order to prevent future glycemic decompensation.

ELIGIBILITY:
Inclusion Criteria:

* 36 Obese AA subjects with DKA or severe hyperglycemia and 8 obese nondiabetic subjects, age 19-65. All studies will be performed in the GCRC at Grady Memorial Hospital.
* Subjects with a BMI ≥ 28 kg/m2 will be included.
* Diagnostic criteria for DKA will include:

  * a plasma glucose > 250 mg/dl,
  * a venous pH < 7.30,
  * a serum bicarbonate < 18 mEq/l, and
  * high serum ketones.
* Obese hyperglycemic patients will have:

  * a blood glucose on admission > 400 mg/dl,
  * a serum bicarbonate > 18 mEq/l, and
  * negative ketones.

Exclusion Criteria:

* Patients with significant medical or surgical illness, including but not limited to myocardial ischemia, congestive heart failure, chronic renal insufficiency, liver failure, and infectious processes;
* Patients with recognized endocrine disorders, such as hypercortisolism, acromegaly, or hyperthyroidism;
* Bleeding disorders, or abnormalities in coagulation studies;
* Pregnancy.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 36 Obese AA subjects with DKA or severe hyperglycemia and 8 obese nondiabetic subjects, age 19-65.
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn D Smiley, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Vellanki P, Stefanovski D, Anzola II, Smiley DD, Peng L, Umpierrez GE. Long-term changes in carbohydrate tolerance, insulin secretion and action in African-American patients with obesity and history of hyperglycemic crises. BMJ Open Diabetes Res Care. 2020 May;8(1):e001062. doi: 10.1136/bmjdrc-2019-001062. PMID 32475838